## TGI ICU Power Analysis – FMER Correction 06/25/24

Embedded Palliative Care in the Medical Intensive Care Unit: Power Analysis

Document Upload Date: August 19, 2024

Study Protocol Number: 202406143

Power Analysis Last Updated June 25, 2024

## TGI ICU Power Analysis – FMER Correction 06/25/24

Design: Stepped-wedge design, cross-sectional sampling, exchangeable correlation structure, no varying cluster sizes, 2 steps, 1 cluster per sequence

| С | Period 1 | Period 2 | Period 3 |
|---|----------|----------|----------|
| 1 | 0 | 1 | 1 |
| 2 | 0 | 0 | 1 |

Assumptions: Continuous outcome type, 80% power, .25 effect size, .03 ICC, .025 alpha



438 per cluster (2), per period (3) 876 per period (3) 2628 total for study

## TGI ICU Power Analysis – FMER Correction 06/25/24

Design: Stepped-wedge design, cross-sectional sampling, exchangeable correlation structure, no varying cluster sizes, 2 steps, 1 cluster per sequence

| С | Period 1 | Period 2 | Period 3 |
|---|----------|----------|----------|
| 1 | 0 | 1 | 1 |
| 2 | 0 | 0 | 1 |

Assumptions: Continuous outcome type, 80% power, .20 effect size, .03 ICC, .025 alpha



688 per cluster (2), per period (3) 1376 per period (3) 4128 total for study